CLINICAL TRIAL: NCT00893815
Title: Prevalence and Predictors of Neurocognitive Impairment Among HIV-infected Patients
Status: Completed | Type: Observational
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: Infectious Diseases Clinical Research Program (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); University of California, San Diego (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: IDCRP-016; Y1-AI-5072 (Other Grant/Funding Number: NIAID Interagency Agreement); P30MH062512 (NIH)
Record Dates: First submitted 2009-05-04; First posted 2009-05-06 (Estimated); Results first posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: HIV Infections; Memory
Keywords: HIV; Neurocognitive function
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- 1: HIV-Positive and Early HIV infection (<6 years of HIV infection since diagnosis [based on DoD standard testing], no prior AIDS-defining condition, and CD4 nadir >200 cells/mm3)
- 2: HIV-Positive and Late HIV-infection (HIV infected, not meeting all 3 criteria)
- 3: HIV-negative (HIV uninfected based on DoD standard testing)

SUMMARY:
Despite the advent of highly active antiretroviral therapy (HAART), the prevalence of neurocognitive impairment among HIV-infected patients continues to be an important issue. Although severe forms of AIDS-related dementia have diminished, milder forms of cognitive impairment have been noted among approximately 30% of asymptomatic HIV patients. Studies among HIV-infected U.S. military personnel regarding neurocognitive function have largely been limited to the early 1990s, before the advent of HAART. In these studies subtle neurobehavioral changes were noted among asymptomatic HIV-positive military personnel.

This study proposes to determine the prevalence of neurocognitive deficits among HIV-positive military beneficiaries during the era of HAART who are participants of the U.S. Military HIV Natural History Study. The prevalence ascertained in this study will be compared to HIV-negative military beneficiaries who are demographically similar to the HIV positive group. The sample size of the study is to have complete testing on 200 HIV positive and 50 HIV-negative participants; due to the possibility of attrition before study completion, the investigators will enroll up to 300 participants (240 HIV-positive and 60 HIV-negative) to achieve this sample size. The investigators' rates among HIV-positive patients found in this study will also be contextualized in the setting of the prevalence of prior neurocognitive deficits seen in a HIV positive U.S. military population studied in the 1990s, contemporary rates among civilian HIV-infected persons, and normative values in the general HIV-negative population. Compared to other data in the field of neuropsychology, this study is novel in that the HIV population studied is composed largely of HIV patients who have been diagnosed early in their HIV infection; have open, free access to antiretrovirals to begin therapy earlier than most other cohorts; and consists of highly-functioning, educated individuals.

DETAILED DESCRIPTION:
Abbreviations:

DOD - U.S. Department of Defense; CD4 - cluster of differentiation 4

ELIGIBILITY:
HIV Positive Group:

Inclusion Criteria:

* HIV-infected patients who are 18-50 years of age
* Current participants in the U.S. Military HIV Natural History Study (RV168)

Exclusion Criteria:

* Current suicidal ideation
* Inability or unwillingness to complete the full or abbreviated neuropsychological battery and other questionnaires
* An acute medical condition that may impact the participant's ability to complete the tests or that may have a significant impact on the test results as deemed by the site research physicians (e.g., pneumonia, influenza); the subject may participate at a later date if the physician deems that the acute medical illness is resolved.

HIV Negative Group:

Inclusion Criteria:

* Between 18 and 50 years of age.
* A military beneficiary
* HIV negative by an ELISA drawn within one year of study enrollment (or willingness to have HIV test performed which has a negative result)

Exclusion Criteria:

* Inability or unwillingness to complete the full or abbreviated neuropsychological battery and other questionnaires
* Presence of current suicidal thoughts
* An acute medical condition that may impact the participant's ability to complete the tests or that may have a significant impact on the test results as deemed by the site research physicians (e.g., pneumonia, influenza); the subject may participate at a later date if the physician deems that the acute medical illness is resolved.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population will consist of 50 HIV-negative patients and at least 200 HIV-positive patients who are 18-50 years of age and current participants of "A Retrospective and Prospective Observational Study of the Natural History of HIV Infection in Active Duty U.S. Military Personnel and Department of Defense Beneficiaries"(RV168).
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2009-04 (Actual); Primary Completion 2011-06 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian K Agan, MD, Principal Investigator — Infectious Disease Clinical Research Program (IDCRP)
Locations (3):
- United States (3):
  - Naval Medical Center San Diego, San Diego, California
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Brooke Army Medical Center, Fort Sam Houston, Texas

REFERENCES:
- [Result] Moore DJ, Roediger MJ, Eberly LE, Blackstone K, Hale B, Weintrob A, Ganesan A, Agan BK, Letendre SL, Crum-Cianflone NF. Identification of an abbreviated test battery for detection of HIV-associated neurocognitive impairment in an early-managed HIV-infected cohort. PLoS One. 2012;7(11):e47310. doi: 10.1371/journal.pone.0047310. Epub 2012 Nov 8. PMID 23144815
- [Result] Crum-Cianflone NF, Moore DJ, Letendre S, Poehlman Roediger M, Eberly L, Weintrob A, Ganesan A, Johnson E, Del Rosario R, Agan BK, Hale BR. Low prevalence of neurocognitive impairment in early diagnosed and managed HIV-infected persons. Neurology. 2013 Jan 22;80(4):371-9. doi: 10.1212/WNL.0b013e31827f0776. Epub 2013 Jan 9. PMID 23303852
- [Result] Crum-Cianflone NF, Roediger MP, Moore DJ, Hale B, Weintrob A, Ganesan A, Eberly LE, Johnson E, Agan BK, Letendre S. Prevalence and factors associated with sleep disturbances among early-treated HIV-infected persons. Clin Infect Dis. 2012 May;54(10):1485-94. doi: 10.1093/cid/cis192. Epub 2012 Mar 19. PMID 22431801

RESULTS

PARTICIPANT FLOW:
Groups:
- HIV-Positive and Early HIV Infection: <6 years of HIV infection since diagnosis, no prior AIDS-defining condition, and CD4 count nadir > 200 cells/mm3
- HIV-Positive and Late HIV-infection: >6 years of HIV infection since diagnosis, prior AIDS-defining condition, or CD4 count nadir < 200 cells/mm3
- HIV-negative: HIV-negative, control group
Period: Overall Study
Arm/Group | HIV-Positive and Early HIV Infection | HIV-Positive and Late HIV-infection | HIV-negative
Started | 100 | 100 | 50
Completed | 100 | 100 | 50
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HIV-Positive and Early HIV Infection | HIV-Positive and Late HIV-infection | HIV-negative | Total
Number analyzed (Participants) | 100 | 100 | 50 | 250
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 100 | 100 | 50 | 250
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 28.8 [25.6 to 35.9] | 42.1 [36.9 to 46.5] | 36.0 [27.0 to 44.0] | 36.4 [27.6 to 43.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 2 | 11
  Male | 97 | 94 | 48 | 239
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 44 | 53 | 25 | 122
  Black | 27 | 31 | 4 | 62
  Hispanic | 17 | 11 | 9 | 37
  Other | 12 | 5 | 12 | 29
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 100 | 100 | 50 | 250

OUTCOME MEASURES:

1. Primary Outcome: The Prevalence of Neurocognitive Deficits Among HIV-positive Patients as Defined by the Global Deficit Score Based on the Neuropsychological Testing Battery and to Compare This Rate to HIV-negative Military Personnel.
Description: All participants underwent a comprehensive battery of standardized neuropsychological test and questionnaires that have been shown to be sensitive to HIV-associated neurocognitive disorders. Neuropsychological test were scored by trained psychometrists. Raw scores were converted to demographically adjusted t scores corrected for effects of age, education, gender, and ethnicity. Scores were then converted to deficit scores that give differential weight to impair rather than normal scores. The Global Deficit score was used to summarize neuropsychological test results by quantifying the number and degree of impaired performances. A score of of ≥0.5 has been shown to be a sensitive and specific indicator of global neurocognitive impairment.
Time Frame: within 30 days
Population: To highlight HIV-positive to HIV-negative comparison, HIV-Positive early and late groups were combined in the paper for statistical analyses. Data are presented here in disaggregated form.
Measure: Number (95% Confidence Interval); unit: percentage with Impairment
Groups:
- HIV-Positive-Early: Early HIV infection Participants
- HIV-Positive-Later: HIV positive later stage group
Arm/Group | HIV-Positive-Early | HIV-Positive-Later | HIV-negative
Number analyzed (Participants) | 100 | 100 | 50
percentage with Impairment | 18 [10 to 26] | 20 [12 to 28] | 30 [17 to 43]
Statistical Analysis 1: Comparison: HIV-Positive-Early vs HIV-negative; Test type: Other; p = 0.09, Regression, Logistic — Threshold for statistical significance: 0.05; Odds Ratio (OR) = 0.55, 95% CI 2-sided [0.27 to 1.10] — HIV-positive / HIV-negative

2. Secondary Outcome: The Prevalence of Neurocognitive Impairment Among HIV-positive Compared to HIV-negative Military Beneficiaries in Seven Major Ability Areas.
Description: All participants underwent a comprehensive battery of standardized neuropsychological tests and questionnaires that have been shown to be sensitive to HIV-associated neurocognitive disorders. Neuropsychological tests were scored by trained psychometrists. Raw scores were converted to demographically adjusted t scores corrected for effects of age, education, gender, and ethnicity. Score were then converted to deficit scores that give differential weight to impaired rather than normal scores. The Global Deficit score was used to summarize neuropsychological test results by quantifying the number and degree of impaired performances. A score of ≥0.5 has been shown to be a sensitive and specific indicator of global neurocognitive impairment.
Time Frame: within 30 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- HIV-Positive-Early: Early HIV infection Participants (<6 years of HIV infection since diagnosis, no prior AIDS-defining condition, and CD4 nadir >200 cells/mm3)
- HIV-Positive-Later: Later HIV positive participants (not meeting all 3 criteria for Early stage)
Arm/Group | HIV-Positive-Early | HIV-Positive-Later | HIV-negative
Number analyzed (Participants) | 100 | 100 | 50
Participants
  Verbal Fluency | 15 | 20 | 11
  Abstraction Executive Functioning | 19 | 19 | 12
  Speed of Information Processing | 10 | 7 | 3
  Attention/Working Memory | 23 | 22 | 9
  Learning | 17 | 25 | 19
  Recall | 18 | 19 | 7
  Motor Speed & Dexterity | 25 | 19 | 12
Statistical Analysis 1: Comparison: HIV-Positive-Early vs HIV-negative; Comparing prevalence of verbal fluency impairment between HIV-positive and HIV-negative military beneficiaries; Test type: Other; p = 0.45, Regression, Logistic — Threshold for statistical significance: 0.05; Odds Ratio (OR) = 0.75, 95% CI 2-sided [0.35 to 1.61] — HIV-positive / HIV-negative
Statistical Analysis 2: Comparison: HIV-Positive-Early vs HIV-negative; Comparing prevalence of abstraction executive functioning impairment between HIV-positive and HIV-negative military beneficiaries; Test type: Other; p = 0.43, Regression, Logistic — Threshold for statistical significance: 0.05; Odds Ratio (OR) = 0.74, 95% CI 2-sided [0.35 to 1.56] — HIV-positive / HIV-negative
Statistical Analysis 3: Comparison: HIV-Positive-Early vs HIV-negative; Comparing prevalence of speed of information processing impairment between HIV-positive and HIV-negative military beneficiaries; Test type: Other; p = 0.56, Regression, Logistic — Threshold for statistical significance: 0.05; Odds Ratio (OR) = 1.45, 95% CI 2-sided [0.41 to 5.17] — HIV-positive / HIV-negative
Statistical Analysis 4: Comparison: HIV-Positive-Early vs HIV-negative; Comparing prevalence of attention/working memory impairment between HIV-positive and HIV-negative military beneficiaries; Test type: Other; p = 0.49, Regression, Logistic — Threshold for statistical significance: 0.05; Odds Ratio (OR) = 1.32, 95% CI 2-sided [0.60 to 2.93] — HIV-positive / HIV-negative
Statistical Analysis 5: Comparison: HIV-Positive-Early vs HIV-negative; Comparing prevalence of learning impairment between HIV-positive and HIV-negative military beneficiaries; Test type: Other; p = 0.01, Regression, Logistic — Threshold for statistical significance: 0.05; Odds Ratio (OR) = 0.43, 95% CI 2-sided [0.22 to 0.84] — HIV-positive / HIV-negative
Statistical Analysis 6: Comparison: HIV-Positive-Early vs HIV-negative; Comparing prevalence of recall impairment between HIV-positive and HIV-negative military beneficiaries; Test type: Other; p = 0.46, Regression, Logistic — Threshold for statistical significance: 0.05; Odds Ratio (OR) = 1.39, 95% CI 2-sided [0.58 to 3.34] — HIV-positive / HIV-negative
Statistical Analysis 7: Comparison: HIV-Positive-Early vs HIV-negative; Comparing prevalence of motor speed & dexterity impairment between HIV-positive and HIV-negative military beneficiaries; Test type: Other; p = 0.76, Regression, Logistic — Threshold for statistical significance: 0.05; Odds Ratio (OR) = 0.89, 95% CI 2-sided [0.43 to 1.85] — HIV-positive / HIV-negative

ADVERSE EVENTS:
Time Frame: Adverse events were reviewed during active participation in the study (30 days)
Groups:
- HIV-Positive and Late HIV-infection: >6 years of HIV infection since diagnosis, prior AIDS-defining condition, and CD4 count nadir < 200 cells/mm3
Arm/Group | HIV-Positive and Early HIV Infection | HIV-Positive and Late HIV-infection | HIV-negative
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/100 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/100 | 0/50
Other Adverse Events (participants affected / at risk) | 0/100 | 0/100 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No